CLINICAL TRIAL: NCT06506253
Title: Massage for GAD: Neuroimaging and Clinical Correlates of Response
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Mark Rapaport, MD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00153327
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Generalized Anxiety Disorder
Keywords: fMRI; massage; touch
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: This is a two-arm, randomized, single masked study investigating the effects of Swedish massage therapy (SMT) vs. a light touch (LT) control on brain activity, clinical response, and autonomic function in subjects with GAD.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Of necessity, the coordinator, subjects, and therapists will know their randomized group assignment. Other study staff interacting with participants, including the investigator completing adverse event assessments, will be masked to the treatment assignment. Participants randomized to a treatment arm will be asked not to disclose their assigned treatment to those staff members. The study coordinator and therapists performing the SMT and LT interventions will not discuss subjects' treatment assignment with other staff at any time during the study. The study statistician will perform and report the primary and secondary outcome analyses using masked treatment codes. The non-masked coordinator will have access to the study randomization schedule and may unmask subjects only in the case of emergency, or if necessary, to establish proper follow-up treatment for a condition that arises during the course of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Swedish Massage Therapy (Experimental): The therapist uses non-aromatic cream to facilitate making long strokes over the body. Swedish massage is done with the subject covered by a sheet, a technique called "draping." One part of the body is uncovered, massaged, and then re-draped before moving to another part. The primary techniques used in the research protocol therapy are effleurage, petrissage, kneading, tapotement and thumb friction. These techniques are performed in a very precise, carefully elaborated manner. The session starts with the subject fully draped in a prone position on the massage table and after approximately 22 minutes the subject is instructed to turn to the supine position. Finally, the therapist moves to the head area of the subject, begins working on the shoulders, neck and head using effleurage and thumb friction, and concludes by using light tapotement on the head. The total time for the entire massage is 45 minutes. Subjects randomized to SMT will undergo 2/week for a total of 6 weeks.
  Interventions: Other: Swedish Massage Therapy
- Light Touch Control (Active Comparator): The Light Touch Control protocol entails the same duration and sequence of procedures as the massage protocol, except that the therapist employs only light-touch hand placement on the subject's body. This condition isolates the effect of the mechanical intervention of SMT. Subjects randomized to LT will undergo 2/week for a total of 6 weeks.
  Interventions: Other: Light Touch Therapy

INTERVENTIONS:
Other: Swedish Massage Therapy — Touch therapy
  Arms: Swedish Massage Therapy
Other: Light Touch Therapy — Touch therapy
  Arms: Light Touch Control

SUMMARY:
This clinical trial will compare the effects of Swedish massage or light touch therapy on brain activity and symptoms of anxiety.

This is a randomized research study and subjects will be randomized into one of two study touch intervention groups, and will have an equal chance of being placed in one of the groups:

1. Swedish massage therapy twice per week for 6 weeks.
2. Light touch therapy twice per week for 6 weeks.

The Primary Objective is to identify brain networks activated by touch interventions using fMRI brain imaging in subjects with generalized anxiety disorder.

Subjects will undergo two fMRI scanning sessions (one before and one after) twice per week for 6 weeks of touch intervention. Subjects will also be asked to complete questionnaires on anxiety, stress and depression.

DETAILED DESCRIPTION:
This is a two-arm, randomized, single masked study investigating the effects of Swedish massage therapy (SMT) vs. a light touch (LT) control on brain activity, clinical response, and autonomic function in subjects with Generalized Anxiety Disorder (GAD).

Primary Objective:

To identify brain networks activated by SMT vs. LT using resting state fMRI and Functional Connectivity during the fearful faces task in subjects with GAD. Primary endpoint: Pre-to-post-treatment change in resting state functional connectivity.

Secondary Objectives:

To correlate pre-to-post-treatment change in rsFC with changes in anxiety scores (HAM-A) within both treatment groups. Secondary Endpoints: Pre-to-post-treatment change in response to fearful/angry faces task and clinical response on the HAM-A.

To correlate changes in autonomic measures with clinical response and rsFC. Secondary Endpoint: Autonomic activity (heart rate variability, heart rate, pulse).

Exploratory Objectives: To evaluate whether SMT improves stress depression and global functioning more than LT. Exploratory Endpoints: Change in Perceived Stress (Perceived Stress Scale), depression (Quick Inventory of Depressive Symptomatology (QIDS-SR)), and global functioning (Clinical Global Impression-S/I) from baseline to post intervention at week 6.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 18 and < 65 years old.
2. Medically stable.
3. Primary Diagnosis of GAD.
4. Hamilton Rating Scale for Anxiety (HAM-A) ≥15
5. Off concurrent psychotropic medication for at least 2 weeks prior to initiation of randomized treatment, OR stable on current medication for a minimum of 6 weeks (prior to initiation of randomized treatment) and willing to maintain a stable dose.
6. Ability to lie prone or supine for one hour at a time, given the nature of the massage intervention
7. Subjects must have a permanent domicile
8. Subjects must be able to comply with the research protocol
9. Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

1. Current (within 3 months of screening visit) nicotine use, illicit drug use, regular or long-term medication use that, in the opinion of the investigator, could alter the results of the study
2. Pregnancy (per participant report, pregnancy testing not done for study)
3. Usually is asleep during the daytime (ie. due to working third-shift), or any other behaviors that routinely disrupt normal diurnal (daily) rhythms
4. Current (past month) rigorous dieting (defined as <1200 calories per day for ≥2 consecutive days)
5. In the month before screening visit, excessive regular use of alcohol, as defined by either of the following, twice a month or more often: (a drink is one 5 ounce glass of wine or equivalent)

   1. ingestion of 5 drinks or more in a 2 hour period
   2. ingestion of 7 drinks or more in a 24 hour period
6. Initiation of psychotherapy or CAM interventions because of psychological distress within 90 days before screening visit.
7. Has a lifetime diagnosis of PTSD, bipolar disorder, OCD, psychotic disorders, OR a current diagnosis of an alcohol or substance use disorder
8. Meets criteria for current suicidal or homicidal ideation
9. Subjects who have massages on a regular basis. Regular massage usage will be defined as receiving on average 4 or more massages/year for the last 5 years
10. Subjects currently employing any other CAM manual therapy and/or holistic therapies to treat a perceived health problem
11. History of head injury or neurological disorder, that in the investigator's opinion would impact the data or preclude safe and successful completion of the study.
12. History of cancer that required chemotherapy and/or radiation treatment.
13. General contraindication to MRI - Because MRI uses a very strong magnet, subjects cannot have metals in their bodies or certain medical conditions. Subjects cannot have a cardiac pacemaker; hearing aid; any other implant metal in their body or eyes, including pins, screws, shrapnel, plates, teeth braces, or dentures. Subjects cannot have tattoos on their head, such as eyeliner or other permanent makeup, as they may make it impossible to get clear and usable images.
14. Medical, psychiatric, cognitive, or other conditions that may compromise the subject's ability to understand the subject information, give informed consent, comply with the study protocol, or complete the study.
15. Current participation in another research study (excluding large natural cohort trials such as 'All of Us')

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Pre-to-post-treatment change in resting state functional connectivity | 6 weeks
  Identification of brain networks activated by SMT vs. LT using resting state fMRI and Functional Connectivity during the fearful faces task in subjects with GAD.

SECONDARY OUTCOMES:
Pre-to-post-treatment change in response to fearful/angry faces task and clinical response on the HAM-A. | 6 weeks
  Correlation of pre-to-post-treatment change in rsFC with changes in anxiety scores (HAM-A) within both treatment groups.
Autonomic activity (heart rate variability, heart rate, pulse). | 6 weeks
  Correlation of changes in autonomic measures with clinical response and rsFC.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rapaport, Principal Investigator — University of Utah
Locations (1):
- Huntsman Mental Health Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
We will maximize the appropriate sharing of scientific data generated from NIH-funded or conducted research, consistent with privacy, security, informed consent, and proprietary issues. Data management and sharing will be addressed in the informed consent process, including communicating with prospective participants how their scientific data are expected to be used and shared. A certificate of confidentiality will be in place.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Following peer-reviewed publication of our results or the end of the funding period (whichever comes first), de-identified materials and data generated in the course of this project will placed in the a repository.
Access Criteria: We will select a data repository that is appropriate for the data generated from the research project. The scientific data will be findable and identifiable, i.e., via a persistent unique identifier (PID) or other standard indexing tools. Shared scientific data will be made accessible in a timely manner for use by the research community and the broader public. Specifically, scientific data will be made accessible as soon as possible, and no later than the time of an associated publication, or the end of the award/support period, whichever comes first. We will consider relevant requirements and expectations (e.g., data repository policies, award record retention requirements, journal policies) as guidance for the minimum time frame scientific data should be made available. However, we will make scientific data available for as long as it is useful for the larger research community, institutions, and/or the broader public.